CLINICAL TRIAL: NCT07278245
Title: Effects of Active Upper-Limb Exoskeleton Training in Simulated Hyper-Gravity on Fine Motor Performance, Brain-Muscle Connectivity, Cardiovascular System and Stress Responses in Real Hyper-Gravity: the EGOS Pilot Study.
Brief Title: Effects of Active Upper-Limb Exoskeleton Training in Simulated Hyper-Gravity on Fine Motor Performance, Brain-Muscle Connectivity, Cardiovascular System and Stress Responses in Real Hyper-Gravity
Acronym: EGOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre National d'Etudes Spatiales (Other Government)
Collaborators: MEDES Institut de Médecine et de Physiologie Spatiales, Toulouse (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 23-318; ID-RCB Number: 2025-A01589-40 (Other: ANSM)
Record Dates: First submitted 2025-11-25; First posted 2025-12-12 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Motor Learning and Physiological Adaptation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Untrained group
- Trained (Experimental): Trained with the exoskeleton
  Interventions: Other: Training with an exoskeleton

INTERVENTIONS:
Other: Training with an exoskeleton — Training to perform an aiming task under simulated hypergravity via an exoskeleton
  Arms: Trained

SUMMARY:
The aim of the study presented here is to assess the effects of exoskeleton training on performance in a real hypergravity situation. In particular, it will analyze fine motor control, autonomic nervous system regulation and metabolic responses. To this end, the study will compare two groups during a pointing exercise in a centrifuge (hypergravity). One group will have been trained to do this exercise using an exoskeleton, while the other will have been familiarized with the task without the exoskeleton. It will assess whether the exoskeleton can be an effective and accessible training tool for astronauts.

ELIGIBILITY:
Inclusion Criteria:

* Maximum weight of 90 kg
* Maximum sitting butt-to-shoulder distance of 70 cm
* Certified as healthy by a comprehensive clinical assessment
* Normal or corrected to normal vision
* Right-handed tested with Edinburgh-Handedness-Inventory-Test (≥6th percentile, on https://www.brainmapping.org/shared/Edinburgh.php)
* Non smokers
* No alcohol or drug dependence, no medical treatment on a regular basis
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC) or a Global Health Insurance Card (GHIC).
* Free of any engagement during the study
* Test subjects must be able to understand and speak English
* Who agreed to take part in the study and signed the informed consent

Exclusion Criteria:

* Left-handed tested with Edinburgh-Handedness-Inventory-Test (<6th percentile)
* Subjects with experience in experiments on a short arm human centrifuge or under real hyper-gravity
* Non-tolerance to the centrifugation
* Any history or presence of clinically relevant chronic disease
* Refusal to give permission to contact his general practitioner,
* Subject who, in the judgment of the investigator, is likely to be non-compliant during the study, or unable to cooperate because of a language problem or poor mental development,
* Subject in the exclusion period of a clinical research,
* Subject who has received more than 6000 Euros within 12 months for being a research subject,
* Subject who cannot be contacted in case of emergency,
* Vulnerable people according to law "Code de la Santé Publique" (L1121-5 to L1121-8)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-10-27 (Actual); Primary Completion 2025-11-27 (Actual); Study Completion 2026-01-27 (Actual)

PRIMARY OUTCOMES:
Task performance (movement accuracy) | From familiarisation sessions (Day 1 to Day 4) to testing day at Day 5.
  Task performance (movement accuracy) is defined as the difference between the position touched on the screen and the position of the displayed target.
  The participants will be required to perform an aiming movement task using their right arm, directed toward a target.The participants will need to point to the center of the displayed target.

CONTACTS AND LOCATIONS:
Locations (1):
- Medes - Imps, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No